CLINICAL TRIAL: NCT06243081
Title: Comparison of Flipped Classroom and Traditional Methods in Basic Life Support Education
Brief Title: The Flipped Classroom Method in Basic Life Support Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nesrin Ogurlu, Lecturer- PhD, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Basic Life Support Training
Record Dates: First submitted 2023-05-15; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Education
Keywords: Skills Training; Flipped Classroom Teaching; Academic Success; Basic Life Support Training

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study. It was planned to divide the students into two groups as experimental and control groups. Simple random sampling method will be used to determine the experimental and control groups. To ensure randomization, each student will be numbered and data sets (experiment and control) will be created.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Flipped Teaching Method Group) (Experimental): Intervention group students will be given skill training with the Flipped Teaching method.
  Interventions: Other: intervention group (Flipped Teaching Method Group)
- Control group (Traditional Method Group) (No Intervention): Control group students will receive skill training with the traditional method. No intervention will be made.

INTERVENTIONS:
Other: intervention group (Flipped Teaching Method Group) — Students will be given skill training with the Flipped Teaching method, which consists of outside and in-class applications.
  Out-of-Class Practice: A Learning Management System-Web-Based Distance Education System will be created for the Flipped Teaching method. Theoretical course topics and skill training videos will be uploaded to the system 7 days before the course day. Students will be able to watch the video tutorials in the number and frequency they want until the day of the lesson. At the end of the lesson, the mini-exam will be uploaded to the system.
  In-class practice: The researcher will come to the lesson prepared for classroom activities such as "question and answer". Theoretical lectures and skill demonstrations will not be made by the researcher. The researcher will only guide the students. Then, the students will be provided to perform the skill under the guidance of the researcher in the clinical skills laboratory.
  Arms: intervention group (Flipped Teaching Method Group)

SUMMARY:
In this study, it was aimed to determine the effect of the Flipped Classroom Teaching Method on student success and skill learning level in Basic Life Support education.

DETAILED DESCRIPTION:
Basic life support (BLS) is a basic practice that increases survival after cardiac arrest and does not require medication. Cardiac arrest may occur due to various reasons. BLS ensures adequate blood flow to the tissues by pumping blood from the heart. BLS can be applied by all healthcare personnel and people trained in this field. The most important factors affecting survival in out-of-hospital cardiac arrests are the timely arrival of the medical team to the scene and basic life support immediately initiated by those who witnessed the arrest.

Today, students mostly consist of Generation Y and Z. People in this generation have an advanced mindset and a rapid process of acquiring information. They are willing to change and always want to be involved in new approaches. People in this generation are defined as a generation that is smart, fond of freedom, fond of technology and knows how to use technology well. For these generations, technology is the symbol of many things in their lives, and it is one of the issues in which generations Y and Z are superior to Generation X. It is stated that these two generations should be supported with student-centered and technology-based activities rather than traditional teaching.

Developing technology offers many options regarding educational environments, methods and tools. Educators who use these options improve educational processes that include information and communication technologies to help students learn. One of these innovations is the "Inverted classroom model".

In general terms, the flipped classroom completely reverses the traditional learning flow and envisages students learning the subject taught by the instructor in the classroom, outside class hours, from materials recorded electronically. It is possible to deepen and reinforce learning by discussing the subject during class hours and doing reinforcing studies. This process is the exact opposite of the traditional classroom model. In the traditional method, the instructor teaches the lesson in the classroom and the student listens passively. In the flipped classroom, students do the listening part of the lesson on their own at home. On the other hand, they practice the difficult and complex upper steps in the classroom with active learning methods and with the guidance of an instructor.

Due to the increasing number of students and resource scarcity in our country, the use of new methods and models in education is a necessity. In a study, it was determined that Generation Z students preferred the flipped classroom teaching method instead of traditional teaching.

In our country, no teaching example of the flipped classroom learning method has been found in Basic Life Support training. However, the requirements and conditions include exploring the implementation and use of new models such as the flipped classroom learning method; It was decided to conduct this research because it was necessary to collect data on whether the application of this learning method was appropriate for the paramedics who will work in the 112 emergency ambulance team to immediately initiate Basic Life Support and apply it consciously and correctly.

ELIGIBILITY:
Inclusion Criteria:

* Students who are in the First and Emergency Aid Program 1st year student

Exclusion Criteria:

* Students who refused to participate in the study Health vocational high school graduate students Students who take course from below

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Measuring Students' Academic Achievement Levels | To be measured at the end of the study (4 weeks later)
  Students in the control and study groups will evaluate theoretical knowledge with the Theoretical Knowledge Evaluation Form prepared in line with the aims and objectives of the course.
Measuring Students' Skill Levels | To be measured at the end of the study (4 weeks later)
  Students will be asked to practice the Basic Life Support skill on a model. Students' Basic Life Support skill performances will be evaluated with the "Basic Life Support Skills Checklist".

CONTACTS AND LOCATIONS:
Overall Officials: NESRİN OĞURLU, Lecturer-PhD, Principal Investigator — Aydın Adnan Menderes University Aydın Vocational School of Health Services; GÜLENGÜN TÜRK, Prof.Dr., Study Director — Aydın Adnan Menderes University Faculty of Nursing, Department of Nursing Fundamentals; MUSTAFA OĞURLU, Prof.Dr., Study Director — Aydın Adnan Menderes University Faculty of Medicine Department of Anesthesia and Reanimation

IPD SHARING:
Plan to Share IPD: Undecided